CLINICAL TRIAL: NCT01187602
Title: A Pilot Study of Short Non-coding RNA Biomarkers of Predisposition to Ovarian Cancer
Brief Title: Short Non-coding RNA Biomarkers of Predisposition to Ovarian Cancer
Acronym: sncRNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Susan Modesitt, MD, MD, University of Virginia
Other Study IDs: 15099
Record Dates: First submitted 2010-08-22; First posted 2010-08-24 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Women at average risk for ovarian cancer: Women at average risk for ovarian cancer (no first degree relatives with breast or ovarian cancer) undergoing gynecologic evaluation at UVA for non-malignant or routine indications.
- Women with ovarian cancer: Women with known or suspected ovarian cancer who are undergoing evaluation and/or treatment at UVA Cancer Center
- Increased risk for ovarian cancer: Women at increased risk of ovarian cancer based on family history, personal history, or genetic factors defined as either BRCA1 or BRCA2 mutations who still retain both fallopian tubes and both ovaries.

SUMMARY:
The purpose of this study is to create new tests to identify biomarkers for ovarian cancer so that a screening test can be developed. For patients who have a diagnosis of ovarian Cancer, researchers will use blood samples before and after treatment to see if disease status can be determined by measuring the amount of biomarker.

DETAILED DESCRIPTION:
Epithelial ovarian cancer is the most lethal female reproductive malignancy, mainly because 80% of tumors have metastasized beyond the ovary at the time of diagnosis. Screening efforts aimed at improved identification of early stage disease have been largely unsuccessful, because of ovarian cancer's propensity for early spread. Our hypothesis is that this obstacle can be circumvented by identifying biomarkers for the precancerous stage of this disease. Since this pre-cancerous stage is currently undetectable, we instead propose to look for biomarkers in women at very high risk for developing ovarian cancer due to genetic mutations. We hypothesize that identification of markers for genetic predisposition to ovarian cancer will also be informative for detection of biological changes that over time lead to sporadic cancers. Given their increasingly recognized role in states of normal and abnormal growth and differentiation, we hypothesize that short non-coding RNAs (sncRNAs) hold significant promise as biomarkers of ovarian cancer predisposition. We will test these hypotheses in two aims. First, we will identify biomarkers for hereditary ovarian cancer risk by comparing serum-derived sncRNAs in women with and without hereditary risk for ovarian cancer. In the second aim we will define serum-derived sncRNAs correlates of ovarian cancer disease status. We will compare sera from ovarian cancer patients at times of highest and lowest disease burden to those of control, cancer-free subjects. Each aim will provide independent, novel, and important information for future investigations. The sncRNAs found to be differentially expressed in both aims will be prioritized for future validation in women under clinical surveillance for hereditary risk of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing medical care at UVA
* Up to date breast cancer screening
* Subjects must fall into one of the following groups:

  * Women at increased risk of ovarian cancer based on family history, personal history, or genetic factors defined as either BRCA1 or BRCA2 mutations who still retain both fallopian tubes and both ovaries.
  * Women at average risk for ovarian cancer
  * Women with known/suspected or recurrent ovarian cancer who are undergoing evaluation and/or treatment at UVA Cancer Center

Exclusion Criteria:

* Subjects with increased risk for ovarian cancer may not have a history of prior malignancy within the last 10 years excluding cervical carcinoma in situ or basal cell carcinoma
* Pregnancy (self reported)

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women in Gynecologic clinics
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2010-08; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Defining sncRNA alterations associated with hereditary predisposition to ovarian cancer | 24 months
  Serum samples will be collected from patients with known BRCA mutations. As a control, we will recruit age-matched women undergoing gynecologic evaluation for benign disease without any personal or family history of cancer. The normal and BRCA mutation groups will be pooled for deep sequencing. Pooled sample short RNAs will be cloned and subjected to deep sequencing and bioinformatic analysis. Validation of 5-10 differentially expressed sncRNAs is performed by quantitative RT-PCR and Northern blots on individual control and high risk samples.
Identification of serum derived sncRNA biomarkers that correlate with disease burden in ovarian cancer. | 24 months
  In this aim pre- and post-remission samples from twenty women with stage III-IV ovarian cancer will be compared to twenty samples from control cancer-free subjects. Methods used will be essentially identical to those described above however, given the opportunity to use each patient as her own control and thus minimized confounders we believe deep sequencing of samples individually will provide better quality data and more robust statistical comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Modesitt, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States